CLINICAL TRIAL: NCT02078752
Title: A FIRST-IN-HUMAN PHASE 1, DOSE ESCALATION, SAFETY AND PHARMACOKINETIC STUDY OF PF-06647263 IN ADULT PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study Of PF-06647263 In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in sponsor prioritization.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7521001
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Neoplasms; Triple-Negative Breast Cancer
Keywords: ADC; PF-06647263; solid tumors; tumors; neoplasm metastasis; TNBC; Triple negative breast cancer
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — PF-06647263

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Part 1 (Experimental)
  Interventions: Drug: PF-06647263

INTERVENTIONS:
Drug: PF-06647263 — Part 1- PF-06647263 will be administered intravenously in either a 21 day cycle or weekly in cohorts of 2 or more patients starting at a dose of 0.015 mg/kg. Increases in dose will continue until MTD is determined.
Drug: PF-06647263 — Part 2- Patients with triple negative breast cancer will be treated at the MTD or Recommended Phase 2 dose selected in Part 1.

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-06647263 in patients with advanced solid tumors in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

DETAILED DESCRIPTION:
The clinical study will include 2 parts. Part 1 will estimate the MTD in dose escalation cohorts in patients with advanced solid tumors for whom no standard therapy is available in order to establish the RP2D. Part 2 will include patients with previously treated metastatic triple negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of solid tumor that is advanced/metastatic and resistant to standard therapy or for whom no standard therapy is available
* Performance Status of 0 or 1
* Adequate bone marrow, kidney, and liver function
* Part 2 includes advanced triple negative breast cancer patients.

Exclusion Criteria:

* Brain metastases requiring steroids
* Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of study treatment start
* Active and clinically significant bacterial, fungal or viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital (BWH), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Hospital / University of Utah, Salt Lake City, Utah
  - Huntsman Cancer Institute-University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Garrido-Laguna I, Krop I, Burris HA 3rd, Hamilton E, Braiteh F, Weise AM, Abu-Khalaf M, Werner TL, Pirie-Shepherd S, Zopf CJ, Lakshminarayanan M, Holland JS, Baffa R, Hong DS. First-in-human, phase I study of PF-06647263, an anti-EFNA4 calicheamicin antibody-drug conjugate, in patients with advanced solid tumors. Int J Cancer. 2019 Oct 1;145(7):1798-1808. doi: 10.1002/ijc.32154. Epub 2019 Feb 23. PMID 30680712
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7521001&StudyName=A%20Study%20Of%20PF-06647263%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06647263 0.01 mg/kg QW (Part 1): Participants received PF-06647263 0.01 mg/kg once weekly (QW) via intravenous (IV) infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.015 mg/kg QW (Part 1): Participants received PF-06647263 0.015 mg/kg once weekly (QW) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.015 mg/kg Q3W (Part 1): Participants received PF-06647263 0.015 mg/kg every 3 weeks (Q3W) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.02 mg/kg QW (Part 1): Participants received PF-06647263 0.02 mg/kg once weekly (QW) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.03 mg/kg Q3W (Part 1): Participants received PF-06647263 0.03 mg/kg every 3 weeks (Q3W) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.05 mg/kg Q3W (Part 1): Participants received PF-06647263 0.05 mg/kg every 3 weeks (Q3W) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.075 mg/kg Q3W (Part 1): Participants received PF-06647263 0.075 mg/kg every 3 weeks (Q3W) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.1 mg/kg Q3W (Part 1): Participants received PF-06647263 0.1 mg/kg every 3 weeks (Q3W) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.134 mg/kg Q3W (Part 1): Participants received PF-06647263 0.134 mg/kg every 3 weeks (Q3W) via IV infusion from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- PF-06647263 0.015 mg/kg QW (Part 2): Participants with triple negative breast cancer (TNBC) regardless of ephrin-A4 (EFNA4) were enrolled in Part 2 of the study when maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) was determined. They received PF-06647263 0.015 mg/kg once weekly (QW) via IV infusion from Cycle 1 Day 1 to the day that the decision was made to discontinue the participants from the study.
Period: Overall Study
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Started | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Completed | 1 | 6 | 1 | 5 | 2 | 5 | 1 | 3 | 2 | 2
Not Completed | 2 | 7 | 1 | 2 | 1 | 4 | 2 | 3 | 0 | 10
Not completed — Death | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 0 | 1
Not completed — Other | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- PF-06647263 0.134 mg/kg QW (Part 1): Participants received PF-06647263 0.134 mg/kg every 3 weeks (Q3W) from Cycle 1 Day 1 until disease progression, patient refusal, unacceptable toxicity occurred or the study was terminated.
- Total: Total of all reporting groups
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2) | Total
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12 | 60
Age, Customized [Count of Participants; unit: Participants]
  18-44 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
  45-64 | 2 | 4 | 2 | 6 | 3 | 9 | 1 | 3 | 0 | 8 | 38
  >=65 | 1 | 7 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 3 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 2 | 7 | 3 | 7 | 2 | 4 | 2 | 12 | 54
  Male | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 11 | 1 | 6 | 3 | 5 | 2 | 6 | 2 | 10 | 48
  Black | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 6
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Unspecified | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) (Part 1)
Description: DLTs were defined as any of the following adverse events (AEs) which were not considered related to disease progression occurring in the first cycle of treatment:(1)Hematologic: grade 4 neutropenia lasting >7 days; febrile neutropenia (defined as neutropenia >=Grade 3 and a single body temperature >38.3°C or a sustained temperature of >=38°C for more than 1 hour); grade >=3 neutropenia with infection; any grade thrombocytopenia associated with clinically significant or life threatening bleeding; grade 4 thrombocytopenia >=72 hours or platelets <=10,000/mm^3 regardless of duration. (2)Non- hematologic: bilirubin increase >=2 × upper limit of normal (ULN) and not related to disease progression or other known cause; all other Grade >=3 toxicities, except those that had not been maximally treated (eg, nausea, vomiting, diarrhea); delay by more than 2 weeks in receiving the next scheduled cycle due to persisting toxicities not attributable to disease progression.
Time Frame: Baseline up to Cycle 2 Day 1 (22 days)
Population: The analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2
Participants | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 2

2. Primary Outcome: Percentage of Participants With Objective Response (Part 2)
Description: Objective response rate (ORR) refers to percentage of participants who achieved complete response (CR) or partial response (PR) determined by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. A participant achieved CR if both target and non-target lesions achieved CR, no new lesions; achieved PR if target lesions achieved CR or PR, non-target lesions were assessed as non-CR/non-PD (progressive disease), indeterminate or missing, and no new lesions. For target lesions, CR: complete disappearance of all target lesions except nodal disease (target nodes must decrease to normal size); PR: >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. For non-target lesions, CR: disappearance of all non-target lesions and normalization of tumor marker levels and all lymph nodes must be normal in size; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: The analysis set included all treated participants in Part 2 with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 12
Percentage of Participants | 8.3 [0.2 to 38.5]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) (All Causality, All Cycles)
Description: An AE was any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Any events occurring following start of treatment or increasing in severity were counted as treatment-emergent.
Time Frame: Baseline up to 28 days after the last treatment administration (Approximately 13 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12

4. Secondary Outcome: Number of Participants With Treatment-Emergent AEs (Treatment-related, All Cycles)
Description: as for outcome 3
Time Frame: Baseline up to 28 days after the last treatment administration (Approximately 13 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Number; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants | 3 | 11 | 2 | 7 | 3 | 9 | 3 | 5 | 2 | 8

5. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (SAEs) (All Causality, All Cycles)
Description: A SAE was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. Any events occurring following start of treatment or increasing in severity were counted as treatment-emergent.
Time Frame: Baseline up to 28 days after the last treatment administration (Approximately 13 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Number; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants | 1 | 6 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 4

6. Secondary Outcome: Number of Participants With Treatment-Emergent SAEs (Treatment-related, All Cycles)
Description: as for outcome 5
Time Frame: Baseline up to 28 days after the last treatment administration (Approximately 13 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Number; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

7. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Following parameters were analyzed for examination of vital signs: sitting systolic and diastolic blood pressure (SBP & DBP), and sitting pulse rate. The abnormal criteria were: (1) minimum SBP <90mmHg; (2) SBP change from baseline, maximum decrease >=30mmHg or maximum increase >=30mmHg; (3) minimum DBP <50mmHg; (4) DBP change from baseline, maximum decrease >=20mmHg or maximum increase >=20mmHg; (5) minimum supine pulse rate <40 BPM or maximum supine pulse rate >120 BPM.
Time Frame: Baseline, Days 1, 8, 15 of each cycle, and post treatment period. (Approximately 13 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants
  Sitting systolic blood pressure (SBP) <90 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  Sitting diastolic blood pressure (DBP) <50 | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 0
  Sitting pulse rate <40 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting pulse rate >120 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
  Max increase from baseline in sitting SBP >=30 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
  Max increase from baseline in sitting DBP >=20 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
  Max decrease from baseline in sitting SBP >=30 | 1 | 5 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 0
  Max decrease from baseline in sitting DBP >=20 | 1 | 3 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0

8. Secondary Outcome: Area Under the Serum Concentration-time Profile From Time 0 to the 504-hour Time Point (AUC504) of PF-06647263
Description: AUC504 was determined by linear/log trapezoidal method. AUC504 analysis only applied to QW groups.
Time Frame: Cycle 1 Day 1: predose, 1, 4, 24, 72 hrs postdose, Cycle 1 Days 8 and 15: predose, 1 and 72 hrs postdose, up to Cycle 2 Day 1 predose (504 hr).
Population: The analysis population was defined as all enrolled patients treated who had sufficient information to estimate AUC504.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 10 | 6 | 8
ng*hr/mL | 2299 (41) | 2777 (26) | 3958 (45) | 3414 (23)

9. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time Tau (AUCtau) of PF-06647263
Description: Tau is dosing interval, where tau=168 hours for the QW dosing and 504-hour for the Q3W dosing. AUC tau was determined by linear/log trapezoidal method. In time frame, C=cycle, D=day.
Time Frame: QW: C1D1: predose, 1,4,24,72 hrs postdose, C1D8 & 15: predose, 1 & 72 hrs postdose, up to C2D1 predose. Q3W: C1D1: predose,1,4 and 24 hrs postdose, C1D4,8,15 up to C2D1 predose; C4D1: pre-dose,1,4 and 24 hrs postdose, C4D4,8,15 up to C5D1 predose.
Population: "Number of Participants Analyzed" represents the number of participants who were enrolled and received at least 1 dose of PF-06647263. "Number Analyzed" represents the number of participants contributing to the PK parameter summary statistics at that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 11 | 2 | 6 | 3 | 5 | 3 | 4 | 2 | 12
  Cycle 1 Day 1 | 594.1 (38) | 544.8 (28) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were :458 and 1360 | 1056 (31) | 1246 (56) | 3475 (36) | 6023 (35) | 6363 (18) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 8060 and 13400 | 669.9 (31)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 9 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 8
  Cycle 1 Day 15 | 927.8 (33) | 1166 (37) |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 1370 and 1570 |  |  |  |  |  | 1274 (30)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 1800 and 1900. | 4617 (42) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 10200. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 6820. |  |

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-06647263
Description: Maximum observed serum concentration Cmax was determined directly from data. In time frame, C=cycle, D=day.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
ng/mL
  Cycle 1 Day 1 | 12.64 (20) | 11.96 (26) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 12.8 and 21.8. | 22.63 (24) | 25.41 (60) | 58.25 (40) | 84.40 (38) | 101.6 (34) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 131 and 154. | 16.86 (29)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 12 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 12
  Cycle 1 Day 15 | 11.86 (33) | 13.73 (47) |  | 27.45 (48) |  |  |  |  |  | 17.84 (25)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 21.2 and 18.1. | 41.98 (16) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 47.7 and 80.9. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 67.7 and 43.8. |  |

11. Secondary Outcome: Time for Cmax (Tmax) of PF-06647963
Description: Tmax was determined directly from data as time of first occurrence. In time frame, C=cycle, D=day.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
hr
  Cycle 1 Day 1 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 4.00] | 2.52 [1.00 to 4.03] | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 1.05] | 1.00 [0.85 to 4.00] | 3.97 [1.05 to 4.05] | 1.05 [1.00 to 1.12] | 1.03 [1.02 to 1.03] | 1.00 [1.00 to 4.00]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 12 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 12
  Cycle 1 Day 15 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] |  | 1.00 [1.00 to 1.00] |  |  |  |  |  | 1.00 [1.00 to 1.00]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | 2.55 [1.00 to 4.10] | 1.08 [1.00 to 4.00] | 2.60 [1.07 to 4.13] | 1.56 [1.05 to 2.07] |  |

12. Secondary Outcome: Clearance (CL) of PF-06647263
Description: For single dose, CL was determined by Dose/AUCinf while for multiple dose, CL was determined by Dose/AUCtau. AUCinf was the area under the serum concentration-time profile from time 0 extrapolated to infinite time. In time frame, C=cycle, D=day.
Time Frame: QW: C1D15: predose, 1 & 72 hrs postdose, up to C2D1 predose. Q3W: C1D1: predose,1,4 and 24 hrs postdose, C1D4,8,15 up to C2D1 predose; C4D1: pre-dose,1,4 and 24 hrs postdose, C4D4,8,15 up to C5D1 predose.
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
L/hr
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 7 | 3 | 5 | 2 | 0
  Cycle 1 Day 1 |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.938. |  | 1.547 (33) | 1.108 (24) | 0.9244 (43) | 0.9219 (39) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 1.06 and 0.807. |
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 9 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 8
  Cycle 1 Day 15 | 0.7932 (15) | 0.9454 (31) |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 0.699 and 0.868. |  |  |  |  |  | 0.8451 (27)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 0.944 and 1.47. | 0.6904 (36) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.441. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.601. |  |

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-06647263
Description: Vss was determined by CL × MRT (mean residence time). MRT=[AUMCtau +tau(AUCinf-AUCtau)]/AUCtau. AUMCtau was the area under the first moment curve derived using the linear/log trapezoidal method. In time frame, C=cycle, D=day.
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
L
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 7 | 3 | 5 | 2 | 0
  Cycle 1 Day 1 |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 116. |  | 162.7 (44) | 114.8 (20) | 134.0 (49) | 116.5 (56) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value were 128 and 159. |
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7
  Cycle 1 Day 15 | 84.01 (28) | 102.3 (49) |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 96.1. |  |  |  |  |  | 72.31 (21)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 123 and 187. | 105.7 (18) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. One of the individual values was 84.6. The other was not reported because CL value did not meet reporting criteria. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. One of the individual values was 109. The other was not reported because CL value did not meet reporting criteria. |  |

14. Secondary Outcome: Terminal Serum Half-life (t1/2) of PF-06647263
Description: T1/2 was determined by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve. The t1/2 analysis only applied to Q3W group. In time frame, C=cycle, D=day.
Time Frame: Q3W: C1D1: predose,1,4 and 24 hrs postdose, C1D4,8,15 up to C2D1 predose; C4D1: pre-dose,1,4 and 24 hrs postdose, C4D4,8,15 up to C5D1 predose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1)
Number analyzed (Participants) | 2 | 3 | 9 | 3 | 6 | 2
day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 7 | 3 | 5 | 2
  Cycle 1 Day 1 | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values.. The individual value was 4.76. | 4.403 (0.593) | 3.541 (0.756) | 5.353 (0.542) | 4.336 (1.02) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value were 5.16 and 5.28.
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 2 | 3 | 2 | 2 | 0
  Cycle 4 Day 1 |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 4.16 and 4.22. | 5.100 (1.56) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 4.93 and 5.79. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 4.77 and 6.07. |

15. Secondary Outcome: AUC504 of Total Antibody
Description: AUC504 was determined by linear/log trapezoidal method. AUC504 analysis only applied to QW groups. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538).
Time Frame: as for outcome 8
Population: The analysis population was defined as all enrolled patients treated who had sufficient information to estimate AUC504.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 11 | 4 | 8
ng*hr/mL | 50080 (38) | 64190 (26) | 91730 (19) | 74250 (40)

16. Secondary Outcome: AUCtau of Total Antibody
Description: Tau is dosing interval, where tau=168 hours for the QW dosing and 504-hour for the Q3W dosing. AUC tau was determined by linear/log trapezoidal method. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538). In time frame, C=cycle, D=day.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 11 | 2 | 6 | 3 | 5 | 3 | 4 | 2 | 11
  Cycle 1 Day 1 | 12140 (29) | 11780 (32) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 10500 and 38500. | 18900 (26) | 38330 (63) | 81710 (45) | 173000 (39) | 164400 (22) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 191000 and 419000. | 13950 (29)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 10 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 7
  Cycle 1 Day 15 | 21620 (30) | 29740 (33) |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 35100 and 35300. |  |  |  |  |  | 32760 (39)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 61500 and 95900. | 155800 (62) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 398000. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 265000. |  |

17. Secondary Outcome: Cmax of Total Antibody
Description: Cmax was determined directly from data. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538). In time frame, C=cycle, D=day.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 8 | 3 | 6 | 2 | 11
  Cycle 1 Day 1 | 209.1 (23) | 187.7 (23) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 240 and 424. | 357.2 (20) | 482.9 (52) | 865.9 (32) | 1475 (45) | 1622 (32) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 2120 and 2860. | 265.3 (27)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 12 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 11
  Cycle 1 Day 15 | 229.6 (25) | 282.7 (32) |  | 506.5 (44) |  |  |  |  |  | 305 (32)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 419 and 462. | 813 (32) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 1170 and 1830. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 1080 and 1320. |  |

18. Secondary Outcome: Tmax of Total Antibody
Description: Tmax was determined directly from data as time of first occurrence. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538). In time frame, C=cycle, D=day.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
hr
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 8 | 3 | 6 | 2 | 11
  Cycle 1 Day 1 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 1.05] | 1.00 [0.850 to 4.00] | 1.05 [1.05 to 4.05] | 1.08 [1.00 to 4.00] | 3.81 [3.62 to 4.00] | 1.00 [1.00 to 4.00]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 12 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 11
  Cycle 1 Day 15 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] |  | 1.00 [1.00 to 1.00] |  |  |  |  |  | 1.00 [1.00 to 72.0]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | 2.55 [1.00 to 4.10] | 1.08 [1.00 to 4.00] | 2.60 [1.07 to 4.13] | 2.55 [1.05 to 4.05] |  |

19. Secondary Outcome: CL of Total Antibody
Description: For single dose, CL was determined by Dose/AUCinf while for multiple dose, CL was determined by Dose/AUCtau. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538). In time frame, C=cycle, D=day.
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
L/hr
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 3 | 0 | 0
  Cycle 1 Day 1 |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.107. |  | 0.04455 (43) | 0.04947 (17) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.0419. | 0.03471 (33) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 10 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 7
  Cycle 1 Day 15 | 0.03411 (5) | 0.03736 (35) |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 0.0312 and 0.0339. |  |  |  |  |  | 0.03447 (48)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 0.0276 and 0.0292. | 0.02049 (45) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.0113. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 0.0155. |  |

20. Secondary Outcome: Vss of Total Antibody
Description: Vss was determined by CL × MRT (mean residence time). MRT=[AUMCtau +tau(AUCinf-AUCtau)]/AUCtau. AUMCtau was the area under the first moment curve derived using the linear/log trapezoidal method. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538). In time frame, C=cycle, D=day.
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
L
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 3 | 0 | 0
  Cycle 1 Day 1 |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 6.30. |  | 10.32 (32) | 10.96 (17) | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 13.3. | 8.074 (51) |  |
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cycle 1 Day 15 | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 4.82 and 5.19. | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. Individual values were 5.09 and 6.45. |  |  |  |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values.. Individual values were 3.87 and 4.06.
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  |  | NA (NA) — Individual values are reported when fewer than 3 participants had report able parameter values. The individual value was 5.33. |  |  |  |

21. Secondary Outcome: t1/2 of Total Antibody
Description: T1/2 was determined by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve. The t1/2 analysis only applied to Q3W group. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538). In time frame, C=cycle, D=day.
Time Frame: as for outcome 14
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1)
Number analyzed (Participants) | 2 | 3 | 9 | 3 | 6 | 2
day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 3 | 3 | 1 | 3 | 0
  Cycle 1 Day 1 | NA (NA) — Fewer than 3 subjects had reportable parameter values. The individual value was 1.88. | 7.860 (0.581) | 7.587 (2.34) | NA (NA) — Fewer than 3 subjects had reportable parameter values. The individual value was 10.1. | 7.713 (1.52) |
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 4 Day 1 |  |  | NA (NA) — Fewer than 3 subjects had reportable parameter values. The individual value was 14.8. |  |  |

22. Secondary Outcome: Cmax of Unconjugated Payload CL-184538
Description: Cmax was determined directly from data. PF-06647263 is an antibody-drug conjugate (ADC) which comprises total antibody (PF-06523432) and unconjugated payload ( CL-184538).
Time Frame: Every Cycle: Days 1, 8, 15. up to end of treatment (Approximately 13 months)
Population: The analysis set was defined as enrolled patients who were analyzed for pharmacokinetics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
ng/mL | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL). | NA (NA) — CL-184538 (unconjugated payload) serum exposure was low with the majority of samples below the limit of quantitation (0.0500 ng/mL).

23. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Following parameters were analyzed for laboratory examination: hematology, blood chemistry, coagulation panel, urinalysis and pregnancy test.
Time Frame: Baseline up to 7 days post end of treatment (Approximately 13 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06647263.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants | 2 | 12 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 11

24. Secondary Outcome: Number of Participants With Positive Antibodies for PF-06647263, Total Antibody (PF-06523432), and Unconjugated Payload (CL-184538)
Description: Positive was defined as: anti-drug antibody (ADA) titer >=1.88. In time frame, C=cycle, D=day.
Time Frame: QW: C1:D1&D15; every other cycle: D1; end of treatment. Q3W:C1: D1&D15; Cycles 2 through 4: D1; every other cycle: D1; end of treatment.
Population: "Number of Participants Analyzed" represents the number of participants who were enrolled and received at least 1 dose of PF-06647263. "Number Analyzed" represents the number of participants tested for that parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants
  Positive Anti-PF-06647263 | 2 | 5 | 0 | 4 | 2 | 4 | 1 | 1 | 0 | 8
  Positive Anti PF-06523432: number analyzed (Participants) | 2 | 5 | 0 | 4 | 2 | 4 | 1 | 1 | 0 | 8
  Positive Anti PF-06523432 | 0 | 3 |  | 0 | 0 | 0 | 0 | 0 |  | 1
  Positive Anti CL-184538: number analyzed (Participants) | 2 | 5 | 0 | 4 | 2 | 4 | 1 | 1 | 0 | 8
  Positive Anti CL-184538 | 2 | 5 |  | 2 | 2 | 4 | 1 | 0 |  | 6

25. Secondary Outcome: Number of Participants With Positive Neutralizing Anti PF-06647263 Antibody
Description: Positive was defined as: neutralizing antibody titer >=1.30. In time frame, C=cycle, D=day.
Time Frame: as for outcome 24
Population: The analysis set included all participants who were treated and tested for that parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 2 | 5 | 0 | 4 | 2 | 4 | 1 | 1 | 0 | 8
Participants | 2 | 5 |  | 3 | 2 | 3 | 1 | 0 |  | 8

26. Secondary Outcome: Number of Participants With Treatment-Emergent and Treatment-Boosted Anti PF-06647263 Antibody
Description: Treatment-Emergent=Baseline negative with at least one positive ADA sample post-treatment. Treatment-Boosted=Baseline positive but endpoint titer (log10-scale titer) increases by at least 0.5 (representing 3-fold titer increase). In time frame, C=cycle, D=day.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 3 | 13 | 2 | 7 | 3 | 9 | 3 | 6 | 2 | 12
Participants
  Treatment-emergent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Treatment-boosted | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Percentage of Participants With Objective Response (Part 1)
Description: as for outcome 2
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: The analysis set included treated participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1)
Number analyzed (Participants) | 2 | 11 | 1 | 6 | 3 | 7 | 3 | 6 | 2
Percentage of participants | 0 [0.0 to 84.2] | 9.1 [0.2 to 41.3] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1] | 0 [0.0 to 70.8] | 14.3 [0.4 to 57.9] | 66.7 [9.4 to 99.2] | 0 [0.0 to 45.9] | 0 [0.0 to 84.2]

28. Secondary Outcome: Percentage of Participants With Clinical Benefit Response
Description: Clinical Benefit Response (CBR) was defined as a CR, PR or stable disease (SD) ≥6 cycles. CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as the reference of baseline sum diameters. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (progressive disease: >=20% increase in the sum of diameters of target lesions and an absolute increase of >=5mm or appearance of >=1 new lesion), taking as reference the smallest sum diameters while on study.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: The analysis set included the number of participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 2 | 11 | 1 | 6 | 3 | 7 | 3 | 6 | 2 | 12
Percentage of participants | 50.0 [1.3 to 98.7] | 36.4 [10.9 to 69.2] | 0 [0.0 to 97.5] | 16.7 [0.4 to 64.1] | 33.3 [0.8 to 90.6] | 42.9 [9.9 to 81.6] | 66.7 [9.4 to 99.2] | 16.7 [0.4 to 64.1] | 0 [0.0 to 84.2] | 25.0 [5.5 to 57.2]

29. Secondary Outcome: Progression Free Survival
Description: The progression free survival (PFS) was defined as the time from Cycle 1 Day 1 to first documentation of disease progression or to death due to any cause, whichever occurred first. PFS was characterized by the estimate median time to event which was derived using Kaplan-Meier method.
Time Frame: Baseline, every 6 weeks until disease progression or unacceptable toxicity up to 24 months
Population: The analysis set included the number of participants with event.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg Q3W (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 0 | 8 | 0 | 4 | 2 | 4 | 1 | 2 | 1 | 8
month |  | 3.0 [1.4 to 7.1] |  | 1.4 [0.6 to 8.3] | 5.3 [1.9 to 5.3] | 5.8 [1.9 to 7.3] | NA [1.4 to NA] — With only one participant, we cannot calculate median or meaningful CI. | 2.8 [0.6 to NA] — Only 33.3% (2/6) of the participants were with event. A 95% CI for the quantile is the set of all efficacy endpoint variable values satisfying the formula. In this group, only one variable value satisfied, so upper limit was not estimable. | NA [1.3 to NA] — With only one participant, we cannot calculate median or meaningful CI. | 1.4 [0.7 to 3.0]

30. Secondary Outcome: Overall Survival (OS)-Stratifying for EFNA4 Expression (Part 2)
Time Frame: Baseline up to 24 months
Population: OS was not estimable since there were fewer number of participants with event.
Arm/Group | PF-06647263 0.015 mg/kg QW (Part 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last treatment administration (Approximately 13 months)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06647263 0.01 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg Q3W (Part 1) | PF-06647263 0.02 mg/kg QW (Part 1) | PF-06647263 0.03 mg/kg Q3W (Part 1) | PF-06647263 0.05 mg/kg Q3W (Part 1) | PF-06647263 0.075 mg/kg Q3W (Part 1) | PF-06647263 0.1 mg/kg Q3W (Part 1) | PF-06647263 0.134 mg/kg QW (Part 1) | PF-06647263 0.015 mg/kg QW (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 4/13 | 0/2 | 0/7 | 0/3 | 1/9 | 0/3 | 1/6 | 0/2 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 6/13 | 0/2 | 0/7 | 1/3 | 1/9 | 1/3 | 3/6 | 1/2 | 4/12
Other Adverse Events (participants affected / at risk) | 3/3 | 13/13 | 2/2 | 7/7 | 3/3 | 9/9 | 3/3 | 6/6 | 2/2 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06647263 0.01 mg/kg QW (Part 1) (N=3) | PF-06647263 0.015 mg/kg QW (Part 1) (N=13) | PF-06647263 0.015 mg/kg Q3W (Part 1) (N=2) | PF-06647263 0.02 mg/kg QW (Part 1) (N=7) | PF-06647263 0.03 mg/kg Q3W (Part 1) (N=3) | PF-06647263 0.05 mg/kg Q3W (Part 1) (N=9) | PF-06647263 0.075 mg/kg Q3W (Part 1) (N=3) | PF-06647263 0.1 mg/kg Q3W (Part 1) (N=6) | PF-06647263 0.134 mg/kg QW (Part 1) (N=2) | PF-06647263 0.015 mg/kg QW (Part 2) (N=12)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06647263 0.01 mg/kg QW (Part 1) (N=3) | PF-06647263 0.015 mg/kg QW (Part 1) (N=13) | PF-06647263 0.015 mg/kg Q3W (Part 1) (N=2) | PF-06647263 0.02 mg/kg QW (Part 1) (N=7) | PF-06647263 0.03 mg/kg Q3W (Part 1) (N=3) | PF-06647263 0.05 mg/kg Q3W (Part 1) (N=9) | PF-06647263 0.075 mg/kg Q3W (Part 1) (N=3) | PF-06647263 0.1 mg/kg Q3W (Part 1) (N=6) | PF-06647263 0.134 mg/kg QW (Part 1) (N=2) | PF-06647263 0.015 mg/kg QW (Part 2) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 3 | 2 | 3 | 1 | 3 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye symptom (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0
Mydriasis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 2 | 3 | 1 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Buccal mucosal roughening (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 5 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 4 | 2 | 2 | 1 | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 9 | 2 | 4 | 3 | 4 | 3 | 3 | 2 | 6
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 1 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 1 | 4 | 1 | 2 | 1 | 2 | 1 | 6
Application site erosion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 10 | 1 | 5 | 2 | 6 | 3 | 4 | 2 | 5
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 5 | 0 | 3 | 1 | 2 | 1 | 2 | 1 | 7
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 3
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 2
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Peritoneal fluid analysis (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 6 | 1 | 4 | 2 | 4 | 3 | 4 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 6 | 0 | 2 | 1 | 1 | 1 | 4 | 2 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail bed tenderness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor's decision (for reasons other than safety) due to which data for few outcome measures was not analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT02078752/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT02078752/SAP_001.pdf